CLINICAL TRIAL: NCT00837577
Title: A Phase III, Randomized, Placebo-controlled, Double-blind Clinical Trial and Subsequent Open-label, Extension Clinical Trial to Study the Efficacy and Safety of Addition of Sitagliptin in Japanese Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Diet/Exercise Therapy and Voglibose Monotherapy
Brief Title: MK0431/ONO-5435 Phase III Clinical Trial -Add-on to Voglibose Study for Patients With Type 2 Diabetes Mellitus (MK0431-104)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-104; 2009_535
Record Dates: First submitted 2009-02-03; First posted 2009-02-05 (Estimated); Results first posted 2011-09-13 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; voglibose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin/Sitagliptin (Experimental)
  Interventions: Drug: Sitagliptin; Drug: Voglibose
- Placebo/Sitagliptin (Experimental)
  Interventions: Drug: Comparator: Placebo; Drug: Sitagliptin; Drug: Voglibose

INTERVENTIONS:
Drug: Comparator: Placebo — Placebo to sitagliptin once daily for 12 weeks (double-blind period)
  Arms: Placebo/Sitagliptin
Drug: Sitagliptin — Sitagliptin/Sitagliptin arm only: Sitagliptin 50 mg once daily orally before breakfast for 12 weeks (double-blind period).
  Both arms: Sitagliptin 50 mg once daily orally before breakfast for 40 weeks (open-label period). The dose of sitagliptin was increased up to 100 mg for participants who had an inadequate response to sitagliptin 50mg after treatment Week 20.
  Other Names: Januvia; MK0431; ONO-5435
Drug: Voglibose — All participants received a stable dose of voglibose, in
  accordance with the package insert, throughout the study.

SUMMARY:
The phase III clinical trial examines the efficacy, safety, and tolerability of the addition of MK0431/ONO-5435 to Japanese patients with type 2 diabetes mellitus (T2DM) who have inadequate glycemic control on diet/exercise therapy and voglibose monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Japanese Patients With Type 2 Diabetes Mellitus, Who Have Inadequate Glycemic Control On Diet/Exercise Therapy And Voglibose Monotherapy

Exclusion Criteria:

* Patients Have A History Of Type 1 Diabetes Mellitus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2009-02-05 (Actual); Primary Completion 2010-08-11 (Actual); Study Completion 2010-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Tajima N, Kadowaki T, Okamoto T, Sato A, Okuyama K, Minamide T, Arjona Ferreira JC. Sitagliptin added to voglibose monotherapy improves glycemic control in patients with type 2 diabetes. J Diabetes Investig. 2013 Nov 27;4(6):595-604. doi: 10.1111/jdi.12116. Epub 2013 Jul 21. PMID 24843714

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin/Sitagliptin: Sitagliptin for 12 weeks (double-blind period) followed by sitagliptin for an additional 40 weeks (open-label period).
- Placebo/Sitagliptin: Placebo for 12 weeks (double-blind period) followed by sitagliptin for 40 weeks (open-label period).
Period: Double-blind Period
Arm/Group | Sitagliptin/Sitagliptin | Placebo/Sitagliptin
Started | 70 | 63
Completed | 68 | 63
Not Completed | 2 | 0
Not completed — Clinical Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Open-label Period
Arm/Group | Sitagliptin/Sitagliptin | Placebo/Sitagliptin
Started | 68 | 63
Completed | 60 | 54
Not Completed | 8 | 9
Not completed — Clinical Adverse Event | 2 | 2
Not completed — Laboratory Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 4 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Other Reason | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin/Sitagliptin | Placebo/Sitagliptin | Total
Number analyzed (Participants) | 70 | 63 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.34 (10.25) | 58.60 (9.73) | 60.57 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 18 | 46
  Male | 42 | 45 | 87
Region of Enrollment [Number; unit: participants]
  Japan | 70 | 63 | 133
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent] | 7.52 (0.75) | 7.50 (0.84) | 7.51 (0.79)
2-hour Postprandial Glucose [Mean (Standard Deviation); unit: mg/dL] | 217.99 (53.22) | 209.40 (52.42) | 213.92 (52.82)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 152.69 (37.06) | 151.54 (30.57) | 152.14 (34.02)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 12
Description: Change from baseline measurement, where the baseline measurement was obtained at randomization (Week 0) before receiving study medication. This study used Japan Diabetes Society (JDS)-certified HbA1c values, the standard at the time when the study was conducted (HbA1c [National Glycohemoglobin Standardization Program; NGSP] = HbA1c (JDS-HbA1c [%]) + 0.4%).
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS) defined as all randomized participants except those participants who did not provide written consent, who were found to be ineligible for the study, or have not taken any study drug during the study period.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of glycosylated hemoglobin
Arm/Group | Sitagliptin/Sitagliptin | Placebo/Sitagliptin
Number analyzed (Participants) | 70 | 63
Percentage of glycosylated hemoglobin | -0.76 (0.42) [-0.88 to -0.63] | 0.16 (0.64) [0.02 to 0.30]
Statistical Analysis 1: Comparison: Sitagliptin/Sitagliptin vs Placebo/Sitagliptin; Test type: Superiority or Other; p < .001, Longitudinal data analysis (LDA) — Adjusted for other prior antihyperglycemic medications (absence, presence); LDA model included both baseline and post-baseline measurements as response variables. P-value calculated using least squares mean; Least squares mean difference = -0.92, 95% CI 2-sided [-1.09 to -0.75], Standard Error of Mean 0.09

2. Secondary Outcome: Change From Baseline in 2-hour Postprandial Glucose at Week 12
Description: Change from baseline measurement, where the baseline measurement was obtained at randomization (Week 0) before receiving study medication.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin/Sitagliptin | Placebo/Sitagliptin
Number analyzed (Participants) | 70 | 63
mg/dL | -55.3 (37.9) [-64.2 to -46.3] | -4.0 (38.7) [-13.5 to 5.5]
Statistical Analysis 1: Comparison: Sitagliptin/Sitagliptin vs Placebo/Sitagliptin; Test type: Superiority or Other; p < .001, Longitudinal data analysis (LDA) — Adjusted for other prior antihyperglycemic medications (absence, presence); [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -51.3, 95% CI 2-sided [-62.3 to -40.2], Standard Error of Mean 5.6

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 12
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin/Sitagliptin | Placebo/Sitagliptin
Number analyzed (Participants) | 70 | 63
mg/dL | -22.6 (27.1) [-28.5 to -16.8] | -0.1 (22.2) [-6.4 to 6.2]
Statistical Analysis 1: Comparison: Sitagliptin/Sitagliptin vs Placebo/Sitagliptin; Test type: Superiority or Other; p < .001, Longitudinal data analysis (LDA) — Adjusted for other prior antihyperglycemic medications (absence, presence); [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -22.5, 95% CI 2-sided [-30.0 to -15.0], Standard Error of Mean 3.8

ADVERSE EVENTS:
Groups:
- Sitagliptin/Sitagliptin (Data Through Week 12): Sitagliptin for 12 weeks (double-blind period) followed by sitagliptin for an additional 40 weeks (open-label period).
- Placebo/Sitagliptin (Data Through Week 12): Placebo for 12 weeks (double-blind period) followed by sitagliptin for 40 weeks (open-label period).
- Pooled Sitagliptin (Data Through Week 52): The Pooled Sitagliptin group includes data from all participants who took sitagliptin in either treatment group: data from Week 0 to Week 52 for participants in the Sitagliptin/Sitagliptin group; data from Weeks 12 through Week 52 for participants in the Placebo/Sitagliptin group; and data from participants in either group who received only sitagliptin 50 mg and those who started on sitagliptin 50 mg and whose dose was subsequently up-titrated to sitagliptin 100 mg orally once daily.
Arm/Group | Sitagliptin/Sitagliptin (Data Through Week 12) | Placebo/Sitagliptin (Data Through Week 12) | Pooled Sitagliptin (Data Through Week 52)
Serious Adverse Events (participants affected / at risk) | 0/70 | 1/63 | 8/133
Other Adverse Events (participants affected / at risk) | 7/70 | 5/63 | 51/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin/Sitagliptin (Data Through Week 12) (N=70) | Placebo/Sitagliptin (Data Through Week 12) (N=63) | Pooled Sitagliptin (Data Through Week 52) (N=133)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Anal Stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin/Sitagliptin (Data Through Week 12) (N=70) | Placebo/Sitagliptin (Data Through Week 12) (N=63) | Pooled Sitagliptin (Data Through Week 52) (N=133)
Nasopharyngitis (Infections and infestations) | 5 (6) | 4 (4) | 40 (66)
Blood Triglycerides Increased (Investigations) | 1 (1) | 0 (0) | 8 (9)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor must have the opportunity to review all communications regarding trial results for 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.